CLINICAL TRIAL: NCT00756340
Title: A Phase I Trial of RAD001 (Everolimus) and Avastin(R) (Bevacizumab) in Children With Recurrent Solid Tumors
Brief Title: A Trial of Everolimus and Bevacizumab in Children With Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RADBEV; NCI-2011-01149 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Recurrent or Refractory Solid Tumors; CNS Malignancies
MeSH Terms: conditions — Recurrence; Central Nervous System Neoplasms | interventions — Bevacizumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): * Dose Level 0, Bevacizumab IV every 2 weeks 8 mg/kg, Everolimus 4 mg/m^2
  * Dose Level 1 (starting dose), Bevacizumab IV every 2 weeks 10 mg/kg, Everolimus 4 mg/m^2
  * Dose Level 2, Bevacizumab IV every 2 weeks 10 mg/kg, Everolimus 5 mg/m^2
  Interventions: Drug: Bevacizumab; Drug: Everolimus

INTERVENTIONS:
Drug: Bevacizumab — * Bevacizumab IV every 2 weeks
  * Dose Level 0- 8 mg/kg
  * Dose Level 1 (starting dose)- 10 mg/kg
  * Dose Level 2- 10 mg/kg
  Other Names: Avastin(R)
Drug: Everolimus — * Everolimus
  * Dose Level 0- 4 mg/m2
  * Dose level 1 (starting dose)- 4 mg/m2
  * Dose Level 2- 5 mg/m2
  Other Names: RAD001; Afinitor(R)

SUMMARY:
The main goals of this Phase I study are to learn about the side effects that may occur when everolimus and bevacizumab are given to children and young adults and to find the highest doses of these drugs that can be given together without causing severe side effects. Bevacizumab will be given into the vein (IV) over 30-90 minutes every two weeks and everolimus tablets will be given daily by mouth. A cycle of therapy will be four weeks.

DETAILED DESCRIPTION:
This is a traditional phase I dose finding study to estimate the maximum tolerated dose (MTD) and describe the dose limiting toxicities (DLT) of the combination of bevacizumab, administered every 2 weeks IV and everolimus administered orally daily to children with recurrent or refractory solid tumors including CNS malignancies. Patients will receive bevacizumab every two weeks IV, and everolimus orally daily. Four consecutive weeks will constitute one course and subsequent courses will immediately follow with no break in the administration of either drug. In the absence of disease progression or unacceptable toxicity, treatment can continue for 2 years. The bevacizumab dose will start at 10 mg/kg. Everolimus will start at 4 mg/m2, 80% of the MTD established in our current phase I trial. A traditional 3+3 dose escalation/de-escalation design will be used to determine the joint MTD for these two agents. Doses to be studied are detailed in the table below. Consistent with the traditional design, we will enroll cohorts of 3 patients at each dose level starting with dose level 1 and will escalate to the next higher dose, if none of these 3 experiences a DLT. If one of 3 patients experiences a DLT at a dose level then 3 more patients will be studied at this level. If none of these 3 experiences a DLT then escalation to the next level will occur. Otherwise the current dose will be considered too toxic and de-escalation will occur. Under this setting, MTD will be the dose level at which 0/3 or 1/6 patient would have experienced DLT and the next dose level is determined to be too toxic.

Exploratory objectives:

1. To preliminarily define the antitumor activity of the combination of everolimus and bevacizumab within the confines of a phase I study
2. To assess the incidence of PTEN and PI3Kinase pathway activation in recurrent or refractory solid tumors of childhood
3. To assess everolimus pharmacokinetics in children, including the effect of concomitant drug therapy (e.g., dexamethasone).
4. To explore changes in correlative magnetic resonance imaging in children receiving everolimus and bevacizumab
5. To identify additional genes both within and outside of the mTOR pathway that may act as determinants of response to everolimus
6. To explore the pharmacogenetic polymorphisms responsible for everolimus disposition (e.g., metabolism and elimination)
7. To test the ability of everolimus to inhibit mTOR pathway signaling in patients with recurrent solid tumors including CNS malignancies in peripheral blood mononuclear cells
8. To estimate blood levels of VEGF, BFGF, TSP-1, I-CAM, v-CAM and circulating endothelial cells prior to, during therapy and after therapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Solid tumor, including central nervous tumors, that is recurrent or refractory to standard therapy or for which standard therapy is not available. All research participants must have a pathologic diagnosis either from their initial presentation, or at the time of recurrence or progression. The requirement for histologic verification may be waived for patients with brainstem glioma and optic pathway glioma.
* Performance Status: Karnofsky > 50% for > 10 years of age; Lansky > 50% for children < 10 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purposes of assessing performance score.
* Neurologic deficits. Patients with CNS tumors must have stable neurological deficits for a minimum of 1 week prior to study entry.
* Life Expectancy: Must be greater than 8 weeks.
* Prior/Concurrent Therapy: Research participants must have recovered from the acute effects of prior treatment and:
* Chemotherapy: Must not have received myelosuppressive chemotherapy within 3 weeks prior to study entry (6 weeks if prior nitrosurea,).
* Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and greater than or equal to 2 months must have elapsed.
* Steroids: Dose should be stable or decreasing for at least one week prior to starting therapy. Corticosteroid therapy is permissible only for the treatment of increased intracranial pressure in patients with malignancies in the CNS or for spinal cord compression. Corticosteroid should be used at the lowest dose to control symptoms and discontinued if possible.
* Must not be receiving tacrolimus or cyclosporine
* Biologic (anti-neoplastic) agent: At least 7 days since the completion of therapy with a biologic agent.
* XRT: Must not have received XRT within 3 months prior to study entry for craniospinal irradiation (>24 Gy) or total body irradiation or if greater than or equal to 50% radiation of pelvis; > 8 weeks for local irradiation to primary tumor; > 2 weeks for focal irradiation for symptomatic metastatic sites.
* Growth factors: Must be off growth factor(s) > 1 week prior to study entry (GCSF, GM CSF, erythropoietin).
* Age: ≤ 21 years.
* Organ Function: Must have adequate organ function and marrow function as defined by the following parameters:
* Bone marrow: peripheral ANC > 1,000/µl, hemoglobin > 8 g/dl (may be transfusion dependent), platelets > 100,000/µ (transfusion independent). (Patients with bone marrow involvement are eligible provided they meet these criteria).
* Hepatic: Bilirubin < 1.5 x institutional upper limit of normal (IULN), SGPT < 3 x IULN.
* Renal: Normal creatinine for age or GFR > 70/ml/min/1.73m2.
* Cardiac: Must have normal EKG and Echocardiogram with shortening fraction > 27% or ejection fraction > 50%.
* Pulmonary: No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% in room air, if there is clinical indication for determination
* Central Nervous System: Patients without seizure disorder OR patients with well-controlled seizure disorder receiving anticonvulsants may be enrolled on this protocol. Anticonvulsants must not be enzyme-inducing (i.e., no barbiturates, phenytoin, carbamazepine, etc, please see Appendix II for a list of drugs that are inducers and inhibitors of CYP3A)
* Informed consent explained to and signed by parent/legal guardian or patient if the patient is ≥ 18 years.
* Patient must begin therapy within 7 calendar days of registration.
* Patient must be able to swallow whole tablets

Exclusion Criteria:

* Concurrently receiving any other concomitant anticancer or experimental drug therapy.
* Have ≥ Grade 2 uncontrolled hypertension
* History of a stroke, myocardial infarction, or unstable angina in the previous 6 months
* Evidence of a bleeding diathesis or PT INR>1.5
* Pre-existing Coagulopathy
* Major surgical procedure(s) within previous 4 weeks prior to study enrollment
* Minor surgical procedures within 7 days prior to study enrollment
* History of an abdominal fistula, GI perforation, or intra-abdominal abscess within previous 6 months.
* A serious, non-healing wound, ulcer, or bone fracture
* In patients with CNS tumors or known CNS metastases, evidence of intracranial or intratumoral hemorrhage on baseline MRI obtained within 14 days prior to study registration.
* If there is proteinuria present on dipstick, patients are excluded if they have >500 mg protein on 24 hour urine collection.
* Require treatment with any of the medications listed in Appendix II (Excluding dexamethasone: Corticosteroid therapy is permissible only for the treatment of increased intracranial pressure in patients with malignancies in the CNS or for spinal cord compression. Corticosteroid should be used at the lowest dose to control symptoms and discontinued if possible).

Use of H2 antagonists such as ranitidine, cimetidine and proton pump blockers such as omeprazole are permissible only in conjunction with corticosteroids in the setting of increased intracranial pressure or for spinal cord compression, as these drugs interfere with CYP3A4. If patients are given such drugs, they must be taken at least 4 hours after intake of everolimus.

* Have an uncontrolled infection.
* History of infection with the hepatitis B and/or C viruses or positive hepatitis B virus surface antigen and hepatitis C virus antibody.
* Pregnant. Females of childbearing potential must have negative serum or urine pregnancy test within 7 days prior to study entry. The effects of everolimus on the developing human fetus are unknown. However, bevacizumab is known to be teratogenic and detrimental to fetal development in animal models. In addition, bevacizumab may alter corpus luteum development and endometrial proliferation, thereby having a negative effect on fertility. For these reasons, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately and will be removed from the study.
* Breastfeeding. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with everolimus or bevacizumab, breastfeeding should be discontinued if the mother is treated on this study.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2008-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To estimate the MTD and describe the DLT of the combination of bevacizumab, administered every 2 weeks IV and everolimus administered orally daily to children with recurrent or refractory solid tumors including CNS malignancies | Within 30 days per subject

CONTACTS AND LOCATIONS:
Overall Officials: Victor Santana, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Santana VM, Sahr N, Tatevossian RG, Jia S, Campagne O, Sykes A, Stewart CF, Furman WL, McGregor LM. A phase 1 trial of everolimus and bevacizumab in children with recurrent solid tumors. Cancer. 2020 Apr 15;126(8):1749-1757. doi: 10.1002/cncr.32722. Epub 2020 Jan 22. PMID 31967673
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols